CLINICAL TRIAL: NCT06806709
Title: Reducing Blood Culture Contamination With the Use of a Needle-less Blood Draw Device (PIVO Pro): An Adaptive Group Sequential Randomized Controlled Trial (The PIVO Trial)
Brief Title: Reducing Blood Culture Contamination With the Use of a Needle-less Blood Draw Device (The PIVO Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IPVA_24.01
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Blood Culture Contamination; Infection
Keywords: PIVO Pro; Reducing blood culture contamination; Needle-less blood draw
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pathology providers will be blinded to the sample collection type. The trial steering committee will remain blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIVO-Pro Intervention arm (Experimental): In the PIVO Pro arm blood culture (BC) sets will also be collected following standard practice, with the addition of PIVO Pro use to draw one BC set from a newly inserted short peripheral intravenous catheter (PIVC). All steps of care will follow standard practice, with use of the PIVO Pro an additional step. Any further BC sets taken at the same time will be collected from a different body location using venepuncture performed as per standard practice. The PIVO Pro BC collection will follow a set procedure, with all steps performed using aseptic technique
  Interventions: Device: PIVO-Pro needle-free blood collection device
- Control arm (No Intervention): In the control arm, all blood culture (BC) sets will be collected using standard practice (typically 1 each for venepuncture/draw from a newly inserted peripheral intravenous catheter).

INTERVENTIONS:
Device: PIVO-Pro needle-free blood collection device — The PIVO™ Pro Needle-free Blood Collection Device advances a flexible flow tube through the intravenous catheter to access optimal blood draw conditions, overcoming traditional hurdles to collect high-quality, reliable blood samples.
  Arms: PIVO-Pro Intervention arm

SUMMARY:
Blood cultures (BCs) are a blood test to look for an infection. Two problems with the sample collection are contamination by germs outside of the blood and not collecting enough blood in the tube, resulting in unusable samples. Many patients requiring a BC also have a peripheral intravenous catheter ("catheter") but these are not normally used for blood sampling. This means that patients receive many painful needles for both catheter insertion and blood sampling. There is a needle-free blood collection device (PIVO Pro) which can be used with a catheter to collect a blood sample.

The goal of the PIVO Trial is to see if using the PIVO Pro for blood culture sample collection will have a lower amount of contamination than the usual method of blood sample collection. Patients 18 and older at 3 emergency departments will be included. Research nurses will look for patients in emergency who need a blood culture sample taken and they will be asked if they want to be involved in the trial. Half of the participants will use the PIVO Pro to take their blood sample and half will have the usual way of collecting blood.

Participants do not have to do anything specifically for the trial. Information about the blood collection and results of the blood culture will be collected from the medical records and recorded for the trial.

DETAILED DESCRIPTION:
The PIVO™ Pro Needle-free Blood Collection Device (Becton, Dickinson and Company; Franklin Lakes) has been available for around a decade and involves advancing a flexible internal flow tube through the patient's Peripheral Intravenous Catheter (PIVC) to access a fresh blood sample beyond the PIVC tip. There is supporting evidence that PIVO is comparable to venepuncture for yielding non-Blood Culture (BC) samples without haemolysis and clotting and with equivalent laboratory values; does not negatively impact PIVC dwell time or replacement rates; decreases preanalytical errors and PIVC replacement; improves the rate and degree of haemolysis in comparison to venepuncture and central line collection; and reduces the prevalence of hospital-onset bacteraemia. However, there are limitations to previous research. Theoretically, for newly inserted PIVCs, the PIVO Pro will bypass a PIVC contaminated on insertion through the skin, to collect a clean blood sample from beyond the tip while also avoiding complications associated with PIVC blood draw. While the PIVO Pro is used in some hospitals as part of standard care, there is a need to confirm results relating to BCs in a randomized controlled trial (RCT).

The aim of this trial is to examine whether use of the PIVO Pro at initial PIVC start, compared to standard practice, decreases BC draw contamination rates.

Based on the aim, the primary objective is to compare the efficacy of the PIVO Pro with initial PIVC start for reducing contaminated BC episodes, to standard practice for BC set draw. 1148 adult participants will be randomised into the trial.

The secondary objectives are to:

1. Compare the effect of the PIVO Pro with initial PIVC start on fill volume of BC bottles, to standard practice for BC set draw.
2. Compare the efficacy of the PIVO Pro with initial PIVC start for improving the overall quality of BC set samples (composite of non-contamination and adequate fill volume), to standard practice for BC set draw.
3. Compare the efficacy of (i) the PIVO Pro (ii) venepuncture, and (iii) draw from initial PIVC start for BC set draw to achieve non-contamination and adequate fill volume
4. Compare the efficacy of the PIVO Pro with initial PIVC start for reducing antibiotic use, to standard practice for BC set draw.

At one hospital site, a sub-study will be conducted to compare PIVC failure outcomes following BC draw with the PIVO Pro with initial PIVC start, to BC set draw directly from a PIVC. The aim of the sub-study is to compare the rate of thrombus development and narrowing of vessel diameter (mm) in those participants that develop PIVC-associated complications versus those participants who do not.

ELIGIBILITY:
Inclusion Criteria:

* Blood culture requested due to suspected bloodstream infection
* Patients receiving a 22 gauge short peripheral intravenous catheter (or larger)

Exclusion Criteria:

* Patients who have already commenced intravenous antimicrobial medications in the emergency department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1148 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood culture draw success without contamination. | Measured at baseline
  Blood culture draw contamination measured as laboratory identification of a common skin commensal in a single blood culture (BC) set in an episode. Should the same common skin commensal be identified by culture in ≥ 2 blood specimens collected on separate occasions (same or consecutive days; e.g., on the same day as the trial BC set/s draw but several hours later) AND the blood cultures are assigned separate specimen numbers, processed individually, and are reported separately in the final laboratory report, the result will be reclassified as being positive (i.e., not contaminated).

SECONDARY OUTCOMES:
Blood culture draw underfill | Measured at baseline
  Inoculation of blood to optimal fill line on bottles or reported by pathology.
Blood culture set quality | Measured at baseline
  Measured as a composite of blood culture non-contamination and adequate fill volume.
Antibiotic use | Within 1 week of baseline.
  Measured as commencement of any antibiotic in response to blood culture results.

CONTACTS AND LOCATIONS:
Overall Officials: Claire Rickard, Principal Investigator — The University of Queensland
Locations (4):
- Australia (4):
  - Caboolture Hospital, Caboolture, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Robina Hospital, Robina, Queensland
  - The Gold Coast University Hospital, Southport, Queensland

IPD SHARING:
Plan to Share IPD: No